CLINICAL TRIAL: NCT01356680
Title: HD17 for Intermediate Stages - Treatment Optimization Trial in the First-Line Treatment of Intermediate Stage Hodgkin Lymphoma
Brief Title: HD17 for Intermediate Stage Hodgkin Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD17
Record Dates: First submitted 2011-05-13; First posted 2011-05-19 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; intermediate stage; PET
MeSH Terms: conditions — Hodgkin Disease | interventions — Bleomycin; Etoposide; Doxorubicin; Cyclophosphamide; Vincristine; Procarbazine; Prednisone; ABVD protocol; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): 2 cycles BEACOPPescalated plus 2 cycles ABVD followed by 30Gy IF-RT irrespective of FDG-PET results after chemotherapy
  Interventions: Drug: BEACOPPescalated (Bleomycin, Etoposide, Adriamycin, Cyclophosphamide, Vincristine, Procarbazine, Prednisone); Drug: ABVD (Adriamycin, Bleomycin, Vinblastine, Dacarbazine); Radiation: 30Gy IF-RT (Involved-Field Radiotherapy)
- Arm B (Experimental): 2 cycles BEACOPPescalated plus 2 cycles ABVD followed by 30Gy IN-RT if FDG-PET is positive after chemotherapy; 2 cycles BEACOPPescalated plus 2 cycles ABVD and treatment stop if FDG-PET is negative after chemotherapy
  Interventions: Drug: BEACOPPescalated (Bleomycin, Etoposide, Adriamycin, Cyclophosphamide, Vincristine, Procarbazine, Prednisone); Drug: ABVD (Adriamycin, Bleomycin, Vinblastine, Dacarbazine); Radiation: 30Gy IN-RT (Involved-Node Radiotherapy)

INTERVENTIONS:
Drug: BEACOPPescalated (Bleomycin, Etoposide, Adriamycin, Cyclophosphamide, Vincristine, Procarbazine, Prednisone)
Drug: ABVD (Adriamycin, Bleomycin, Vinblastine, Dacarbazine)
Radiation: 30Gy IF-RT (Involved-Field Radiotherapy)
  Arms: Arm A
Radiation: 30Gy IN-RT (Involved-Node Radiotherapy)
  Arms: Arm B

SUMMARY:
This study is designed to test the non-inferiority of the experimental arm compared to the standard arm in terms of progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin Lymphoma
* CS I, II with risk factor (stage IIB with risk factor 1 or 2 are not included)
* large mediastinal mass (>1/3 of maximum transverse thorax diameter)
* extranodal involvement
* elevated ESR
* 3 or more involved nodal areas
* written informed consent

Exclusion Criteria:

* Leucocytes <3000/µl
* Platelets < 100000/µl
* Hodgkin Lymphoma as composite lymphoma
* Activity Index (WHO) >2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1100 (Actual)
Dates: Start 2012-01-13 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years
CR rate | 6 months
  Rate of patients achieving a complete remission (CR/CRu) at final restaging after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University of Cologne, German Hodgkin Study Group
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- [Derived] Lommen M, Weindler JJ, Jablonski J, Rosenbrock J, Borchmann P, Behringer K, Roth KS, Ufton D, Dietlein M, Kobe C, Ferdinandus J. Association between metabolic tumor burden and health-related quality of life in patients with classic Hodgkin lymphoma. Eur J Nucl Med Mol Imaging. 2025 Oct 11. doi: 10.1007/s00259-025-07569-5. Online ahead of print. PMID 41074963
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] van Heek L, Weindler J, Gorniak C, Kaul H, Muller H, Mettler J, Baues C, Fuchs M, Borchmann P, Ferdinandus J, Dietlein M, Voltin CA, Kobe C, Roth KS. Prognostic value of baseline metabolic tumor volume (MTV) for forecasting chemotherapy outcome in early-stage unfavorable Hodgkin lymphoma: Data from the phase III HD17 trial. Eur J Haematol. 2023 Dec;111(6):881-887. doi: 10.1111/ejh.14093. Epub 2023 Aug 29. PMID 37644732
- [Derived] Borchmann P, Plutschow A, Kobe C, Greil R, Meissner J, Topp MS, Ostermann H, Dierlamm J, Mohm J, Thiemer J, Sokler M, Kerkhoff A, Ahlborn M, Halbsguth TV, Martin S, Keller U, Balabanov S, Pabst T, Vogelhuber M, Huttmann A, Wilhelm M, Zijlstra JM, Moccia A, Kuhnert G, Brockelmann PJ, von Tresckow B, Fuchs M, Klimm B, Rosenwald A, Eich H, Baues C, Marnitz S, Hallek M, Diehl V, Dietlein M, Engert A. PET-guided omission of radiotherapy in early-stage unfavourable Hodgkin lymphoma (GHSG HD17): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Feb;22(2):223-234. doi: 10.1016/S1470-2045(20)30601-X. PMID 33539742
- [Derived] Voltin CA, Goergen H, Baues C, Fuchs M, Mettler J, Kreissl S, Oertl J, Klaeser B, Moccia A, Drzezga A, Engert A, Borchmann P, Dietlein M, Kobe C. Value of bone marrow biopsy in Hodgkin lymphoma patients staged by FDG PET: results from the German Hodgkin Study Group trials HD16, HD17, and HD18. Ann Oncol. 2018 Sep 1;29(9):1926-1931. doi: 10.1093/annonc/mdy250. PMID 30010775
- See also: Homepage GHSG — http://www.ghsg.org